CLINICAL TRIAL: NCT03274869
Title: Prediction and Early Diagnosis for Cardiovascular Disease Complicated by Scrub Typhus Infection
Brief Title: Scrub Typhus Infection Induced Cardiovascular Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Eulji University Hospital (Other)
Collaborators: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Chungbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Ki-Woon Kang, MD, Professor, Eulji University Hospital
Other Study IDs: EMC 2017-07-006-001
Record Dates: First submitted 2017-09-03; First posted 2017-09-07 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Scrub Typhus; Cardiovascular Complication
Keywords: Scrub typhus; Cardiovascular Complication
MeSH Terms: conditions — Scrub Typhus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — To find novel genotypes of Orientia tsutsugamushi isolated from Scrub typhus infection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Scrub typhus without cardiovascular complications: Any participants with the scrub typhus infection without cardiovascular complication will be enrolled as a positive control group during admission and clinically followed by 1 year after discharge
- Scrub typhus with cardiovascular complication: Any participants with the scrub typhus infection with cardiovascular complication will be enrolled as a comparison group during admission and clinically followed by 1 year after discharge

SUMMARY:
Scrub typhus infection has been considered as seasonal and endemic infectious disorder with benign feature. However, the increasing mortality rate of scrub typhus has been recently reported in Southeast Asia and cause of death could be a fetal complicating cardiovascular disease. Therefore, the association and predictors for scrub typhus induced cardiovascular disease should be investigated to provide a timely and appropriate diagnosis and to reduce the mortality rate of complicated scrub typhus infection. Therefore, investigators prospectively investigate the association and predictors of cardiovascular disease in the participants with scrub typhus infection.

DETAILED DESCRIPTION:
Scrub typhus is a zoonotic disease caused by Orientia tsutsugamushi confined to East Asia including South Korea. It is characterized by fever, headache, rash, and eschar and the majority of patients without complications can recover with an early diagnosis and proper management with antibiotics. However, the increasing mortality rate of scrub typhus has been recently reported in Southeast Asia. Severe complications can be manifested by respiratory distress syndrome, renal failure, hepatic failure, and cardiovascular disease. Especially, cardiovascular complications can lead to cardiogenic shock and sudden cardiac arrest. Therefore, the association and predictors for scrub typhus induced cardiovascular disease should be investigated to provide a timely and appropriate diagnosis and to reduce the mortality rate of complicated scrub typhus infection. Therefore, investigators prospectively investigate the association and predictors of cardiovascular disease in the participants with scrub typhus infection admitted to 3rd referral centers in South Korea.

ELIGIBILITY:
Inclusion Criteria:

* any participants with scrub typhus infection

Exclusion Criteria:

* patients under age of 18
* pregnancy

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Scrub typhus infection without cardiovascular complication Scrub typhus infection with cardiovascular complication
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular Mortality | one year
  Cardiovascular death including sudden cardiac death

SECONDARY OUTCOMES:
Cardiovascular Complications | one year
  Atrial Fibrillation, Acute Heart Failure including acute myocarditis and Ischemic Heart Dease

CONTACTS AND LOCATIONS:
Overall Officials: Hyu Ryung Cho, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (2):
- South Korea (2):
  - Chung-Buk University Hospital, Chungju, Chung Chung Do
  - Chung-Nam University Hospital, Daejeon, Chung Chung Do

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Chin JY, Kang KW, Moon KM, Kim J, Choi YJ. Predictors of acute myocarditis in complicated scrub typhus: an endemic province in the Republic of Korea. Korean J Intern Med. 2018 Mar;33(2):323-330. doi: 10.3904/kjim.2016.303. Epub 2017 Feb 23. PMID 28226202
- [Result] Jang SY, Kang KW, Kim JH, Kim B, Chin JY, Park SH, Choi YJ, Jung KT, Lee SK. New-onset atrial fibrillation predicting for complicating cardiac adverse outcome in scrub typhus infection. Clin Cardiol. 2019 Dec;42(12):1210-1221. doi: 10.1002/clc.23276. Epub 2019 Oct 3. PMID 31580531
- [Result] Kang KW, Hong KW, Lee SK. Identification of novel variants for complicating cardiac disease in the scrub typhus infection using whole genome sequencing. Korean J Intern Med. 2023 Nov;38(6):865-871. doi: 10.3904/kjim.2023.221. Epub 2023 Nov 1. PMID 37939667